CLINICAL TRIAL: NCT05240365
Title: SDF Modified Hall Technique Versus Conventional Pulpotomy for Management of Carious Primary Molars: A Randomized Clinical Trial
Brief Title: SDF Modified Hall Technique Vs. Conventional Pulpotomy for Management of Carious Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sondos Naserallah (Other)
Responsible Party: Sponsor-Investigator, Sondos Naserallah, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDF Modified Hall
Record Dates: First submitted 2021-12-22; First posted 2022-02-15 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-01

CONDITIONS: Deep Carious Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDF modified Hall technique (Experimental): When Hall technique is used an accurate size of PMC is placed without local anesthesia, caries removal, or tooth preparation.
  SDF is applied directly to carious lesions to arrest caries, the technique is noninvasive and relatively painless that could be a good option for treating dental caries in children
  Interventions: Device: SDF modified Hall technique
- Conventional pulpotomy and stainless steel crown (Active Comparator): Amputation of the coronal pulp and treatment of the remaining vital radicular portion with a long term clinically successful medicament. Then using an accurate size of stainless steel crown.
  Interventions: Device: Conventional pulpotomy and stainless steel crown

INTERVENTIONS:
Device: SDF modified Hall technique — * Preparation for Hall technique and selection of the crown.
  * Clinical application of SDF.
  * Cementation of the selected crown.
  Arms: SDF modified Hall technique
Device: Conventional pulpotomy and stainless steel crown — * Teeth will be anesthetized .
  * Rubber dam will be used and high suction in pulpotomy procedure.
  * Cavity outline will be performed by sterile #330 high speed bur using water spray.
  * Caries will be removed by large spoon excavator.
  * pulpal exposure will be occurred then the roof of pulp chamber will be removed by low speed round bur. Hemostasis will be obtained by applying pressure with moist cotton pellet with saline.
  * Teeth will be treated by using sterile cotton pellet with formcresol for three to five min then, remove it.
  * Pulp stumps of will be dressed with reinforced zinc oxide eugenol, IRM®*
  * Tooth Preparation will be done followed by placement of stainless-steel crown
  Arms: Conventional pulpotomy and stainless steel crown

SUMMARY:
Dental caries in primary teeth is considered the most common oral disease of childhood and it has been investigated in many places throughout the world. In most developed countries, the prevalence of early childhood caries (ECC) ranges between 1% and 12%. In less developed countries, however, the prevalence is much higher, exceeding 70%.

Pulpotomy is a clinical procedure usually performed in primary molars with extensive caries, which implies removal of the coronal pulp and preservation of the radicular pulp. It is based on the ability of the remaining pulp tissue to heal after the affected or infected coronal pulp has been surgically removed. Pulpotomy is a technique that is highly dependent on a number of factors, including diagnosis accuracy, caries excavation method, pulp dressing material, final restoration quality and operator experience.

Silver diamine fluoride (SDF) has recently become a non-invasive treatment option, it is fluid-form material used in prevention and treatment of teeth cavities (or caries). SDF has been demonstrated to be useful in arresting caries development after a cavity has formed. In hundreds of studies, the only common side effect of SDF has been black staining surrounding the area. SDF has the ability to stain anything it comes into contact with, including clothing and oral tissues.

Hall technique is a method for management primary molar decay that involves the use of preformed metal crowns (PMCs) to seal decay. This technique may be able to stop or at least reduce caries progression in primary teeth. The process of fitting the crown is quick and non-invasive.

DETAILED DESCRIPTION:
Dental caries is the most common childhood disease and the most common health issue worldwide, despite a half-century of concerted clinical and public health efforts to eliminate it.Untreated caries causes health issues such as pain, poor quality of life, psychosocial suffering, as well as societal burdens such as reduced productivity at work and school.

In order to reduce disease incidence and burden, meet population-level oral health goals, and address patient concerns, oral health education, home hygiene, avoidance of fermentable carbohydrates, consumption of fluoridated water, and access to and utilization of routine dental screenings, examinations, and care are all critical. Caries prevention and treatment strategies that are safe, easy, effective, low-cost, minimally invasive, and amenable to a variety of community settings are desired by dental public health and oral health stakeholders.

One of the traditional methods of managing carious primary molars in children is conventional pulpotomy with stainless steel crowns (SSCs). Recently, other treatments are being used as silver diamine fluoride (SDF) and the Hall technique.

Primary teeth pulpotomy is defined as amputation of the coronal pulp and treatment of the remaining vital radicular portion with a long term clinically successful medicament. An ideal medicament used for pulpotomy should have a bactericidal effect, enhance healing of the radicular pulp tissue and biocompatible then using an accurate size of stainless steel crown.

Hall technique is one of the most common methods for sealing caries in primary molars nowadays. Dr. Norna Hall, a general dentist from Scotland, originally described Hall technique using preformed metal crowns (PMCs) in the literature in 2006. It has very straightforward biological principles. It can protect the primary tooth till shedding and arrest caries. The superficial plaque layer, which is the most essential element in the biofilm for caries growth, is left and sealed together with the carious lesion when using Hall technique. As a result, the plaque biofilm flora will be changed to be less cariogenic that may arrest or reduce the progression of caries in primary teeth.

SDF has been proven to be effective in caries arrest. It's used to manage early childhood caries. Silver and fluoride ions combine to form SDF, a colorless ammonia solution. The fluoride in SDF has a long history of exaggerating enamel and dentine remineralization, while silver has been shown to have potent antimicrobial properties.

ELIGIBILITY:
Inclusion Criteria:

* Children: Age 4 to 7 years medically free.
* Primary molars with deep caries.
* Vital pulp with no clinical signs and symptoms of irreversible pulpitis such as spontaneous pain.
* Absence of swelling or pus exudate or fistula.
* Absence of abnormal teeth mobility
* Absence of pain on percussion

Exclusion criteria:

* Patients experience signs or symptoms of pulpal or periapical pathology.
* Patients requiring special dental consideration.
* Unmotivated uncooperative patients.
* Patients can't attend follow up visits.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours postoperatively
  Any pain and discomfort experienced by the child were recorded using the Faces Pain Scale-Revised (FPS-R).The endpoints were labeled 'no pain' and 'very much pain'. The FPS-R faces were scored as 0-2-4-6-8-10.

SECONDARY OUTCOMES:
Radiographic success | one year
  Obvious furcation or periapical radiolucency by radiographic examination , (Internal and external) resorption by radiographic examination.
Chair side time | immediately after the procedure
  Stop watch (min.s)
Child cooperation | immediately after the procedure
  Evaluate the Child's behavior by Frankl scale (FS) through Scores (1-2-3-4) ,(higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, Professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No